CLINICAL TRIAL: NCT00560534
Title: Whole Body Magnetic Resonance Angiography in Patients With Symptomatic Peripheral Ischemia. Experience With Venous Compression.
Brief Title: Whole Body Magnetic Resonance Angiography With Subsystolic Venous Compression
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Prof. Henrik Thomsen, Copenhagen University Hospital Herlev
Other Study IDs: WB-angio herlev 3
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Atherosclerosis; Intermittent Claudication
Keywords: Magnetic resonance; whole body; angiography; venous compression; MRI
MeSH Terms: conditions — Atherosclerosis; Intermittent Claudication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Whole body magnetic resonance angiography — Magnetic resonance angiography using a paramagnetic contrast agent.Venous compression performed with a blood-pressure cuff around both thighs.

SUMMARY:
To investigate the diagnostic performance of whole body magnetic resonance angiography (WB-MRA) using subsystolic venous compression of the thigh.

DETAILED DESCRIPTION:
WB-MRA is an examination that can evaluate the arteries from head to feet. Timing of the injected bolus of contrast medium can be difficult, especially in the legs. As the result of the WB-MRA depends on the contrast medium only being in the arteries at the time of examination, the use of venous compression is a possible way of overcoming the problem of early venous filling, that can hamper the diagnostic value of the examination. Venous compression is performed with a blod pressure cuff around the thighs. It is inflated to subsystolic pressure (45 mm Hg). This elevated pressure leads to filling of the lower leg arteries and late venous filling.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lower extremity ischemia (claudication, ischemic wounds)
* Referred to digital subtraction angiography (DSA)

Exclusion Criteria:

* Renal insufficiency (GFR < 30 ml/min)
* Contra-indications for MRI-examination (claustrophobia, metal-implants, pacemaker)
* Dementia
* Pregnancy/lactation
* Allergy to gadolinium based MRI contrast agents
* Acute disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2008-06; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Vascular diagnostic quality on the WB-MRA. Degree of arterial stenosis on the WB-MRA | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Henrik S Thomsen, Prof. MD., Study Chair — University Hospital at Herlev Copenhagen Denmark
Locations (1):
- Department of Radiology, Herlev University Hospital, Herlev Copenhagen, Herlev, Denmark